CLINICAL TRIAL: NCT05932004
Title: Does Reformer Pilates Exercise Improve Cognitive Functions in Sedentary Women? A Randomized Controlled Study.
Brief Title: Does Reformer Pilates Exercise Improve Cognitive Functions in Sedentary Women?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Atılım University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-59394181-604.01.02-22602
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Reformer Pilates Exercise, Cognitive Performans

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled study
Who Masked: Participant
Masking Description: Participant will not informed about the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reformer pilates group (Other): Reformer pilates
  Interventions: Other: Reformer pilates exercise
- Control group (Other): intervention waiting group
  Interventions: Other: Reformer pilates exercise

INTERVENTIONS:
Other: Reformer pilates exercise — The reformer Pilates group will receivea 6-week exercise program (45 minutes/twice per week) , while the participants in the control group will be selected from those on the exercise list who will start exercise after the study finishes, but are on a waiting exercise program list

SUMMARY:
The reformer is an apparatus on which to perform the foot work and the body in a comfortable, non weight-bearing supine position and keeps the muscles in balance. Studies on Pilates generally include individuals with chronic diseases, geriatric and obese individuals also active women.

The aim of this study was to investigate the effect of reformer Pilates exercises on cognitive functions in sedentary women

DETAILED DESCRIPTION:
A total of 44 sedentary women aged between 24-50 will be randomized into two groups. The reformer Pilates group will receivea 6-week exercise program (45 minutes/twice per week) , while the participants in the control group will be selected from those on the exercise list who will start exercise after the study finishes, but are on a waiting exercise program list. Outcomes measured before and after the interventions are, right/left discrimination and scores of two questionnaires: Stroop Test and The Pittsburgh Sleep Quality Index.

ELIGIBILITY:
Inclusion Criteria:

* 44 sedentary women aged 25-50 years without regular exercise habits

Exclusion Criteria:

* Individuals who cannot participate to the exercise program regularly,
* those with a serious musculoskeletal or neurological history,
* individuals with communication and emotional problems

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy Sedentary women
Enrollment: 44 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Demographic information | Up to one month
  Demographic information such as age, height, weight, education level and smoking of all individuals participating in the study will be questioned.
Stroop Test | Up to one month
  The Stroop Test Form will be used to evaluate the cognitive functions of the participants such as attention, reaction inhibition, and information processing.
Right-Left Discrimination | Up to one month
  Motor imaging technique left/right discrimination will be used as cognitive evaluation.

SECONDARY OUTCOMES:
Assessment of sleep quality and disorder | Up to one month
  The Pittsburgh Sleep Quality Index will be used to evaluate the sleep quality and disorder of the individuals participating in the study in the past month.

REFERENCES:
- [Derived] Ozeren A, Ulug N, Sahan N, Can Karahan Z. Does reformer pilates exercise improve cognitive functions in sedentary women? A randomized controlled study. J Bodyw Mov Ther. 2024 Oct;40:1899-1905. doi: 10.1016/j.jbmt.2024.10.031. Epub 2024 Oct 18. PMID 39593541